CLINICAL TRIAL: NCT00631085
Title: Effect of Gamma Tocopherol Supplementation on Neutrophil Response to 20,000 EU of Clinical Center Reference Endotoxin in Normal Adults
Acronym: GammaTox
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Michelle Hernandez, MD, UNC_Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GCRC 2678 IRB 08-0082; 5P01AT002620 (NIH)
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Last update posted 2011-04-18 (Estimated); Status verified 2011-04

CONDITIONS: Healthy
Keywords: healthy nonsmoking nonasthmatic volunteers
MeSH Terms: interventions — gamma-Tocopherol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other)
  Interventions: Drug: gamma tocopherol

INTERVENTIONS:
Drug: gamma tocopherol — Maxi Gamma softgels 1200mg QD

SUMMARY:
The purpose of this research study is to learn whether high dose vitamin E (gamma tocopherol) will affect the way your body responds to an acute inflammation in your lungs. Vitamin E is found in soybean and vegetable oils as well as many plant seeds. Gamma tocopherol (gT), a component of vitamin E, composes 70-80% of Vitamin E in the U.S. diet. Alpha tocopherol (aT), another large component of vitamin E, makes up less than 10% of vitamin E in the U.S. diet, but is the major form in blood and tissue. It is also the major form of Vitamin E in over-the-counter supplements. However, gT has anti-inflammatory properties which are not present in aT. Preliminary data suggests that gT protects from ozone-induced exacerbation in animal studies, and previous studies have shown levels of gT are inversely associated with heart disease.

We will ask you to undergo a challenge with endotoxin, which is a bacterial component of air pollution. From other studies we have done, we know that if you inhale 20,000 EUs (endotoxin units) we will see an increase in the number of neutrophils (a type of white blood cell that your body produces to fight infection) in your lung cells without causing you to have flu-like symptoms. We will investigate if there is a change in your lung inflammatory cells after the endotoxin challenge when you take the gT versus when you take a placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy nonsmoking volunteers with normal lung function

Exclusion Criteria:

* Chronic illness
* Asthma
* Active allergies

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2008-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
The primary goal of this study is to determine the effect of γT on endotoxin-induced airway inflammation in non-allergic, non-asthmatic subjects. | CCRE challenge after 7 days of treatment with gT or SO

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, MD, Principal Investigator — University of North Carolina
Locations (1):
- University of North Carolina CEMALB, Chapel Hill, North Carolina, United States